CLINICAL TRIAL: NCT06924515
Title: The Application Value of Intercostal Suturing in Preventing Postoperative Thoracoscopic Lung Resection Chest Wall Pulmonary Hernia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mingjian Ge (Other)
Responsible Party: Sponsor-Investigator, Mingjian Ge, Chief physician;Professor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-491-02
Record Dates: First submitted 2025-04-05; First posted 2025-04-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-04

CONDITIONS: VATS; Lung Hernia
Keywords: lung hernia; VATS

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): After the lung resection-related operations are completed, the chest cavity is properly hemostatic, and the incision protective cover of the relevant operation hole is removed. If there is bleeding in the incision, use electrocoagulation to fully stop the bleeding. After hemostasis is completed, use a ligature suture guide to clamp a 1-0 PDS absorbable suture and insert it into the upper intercostal space on the head side of the main operation port. In the secondary operation space, use a double-jointed separation forceps to grasp the suture in the chest cavity and then detach the suture from the ligature suture guide. At this time, insert the ligature suture guide into the lower intercostal space on the foot side of the main operation port. The suture is clamped by the separation forceps in the chest cavity and then pulled out of the chest cavity after being clamped by the claws of the ligature suture guide. In this way, continuous sutures are performed in sequence for a total of 5 s
  Interventions: Procedure: Intercostal suture
- Control group (No Intervention): After the lung resection operation is completed, the chest cavity is properly hemostatic, and the incision protective cover of the relevant operation hole is removed. If there is bleeding in the incision, electrocoagulation is used to fully stop the bleeding. After the hemostasis is completed, the chest wall muscle group and subcutaneous tissue layer are sutured once with a double-needle barbed suture made of 2-gauge PDO material. Finally, the skin is sutured with ordinary silk thread interrupted sutures or absorbable sutures are used to continuously suture the skin intradermally to complete the chest closure.

INTERVENTIONS:
Procedure: Intercostal suture — 止血完成后使用结扎缝合引线器夹持1-0规格的PDS可吸收缝线在主操作口的头侧上一肋间穿入，于副操作空使用双关节分离钳在胸腔内抓持缝线后将缝线从结扎缝合引线器脱离，此时在主操作口足侧下一肋间穿入结扎缝合引线器，在胸腔内由分离钳夹持缝线经结扎缝合引线器钩爪夹持后将缝线牵拉出胸腔外，以此依次行连续缝合共5次缝合引线操作后拉拢缝线将主操作口闭合，打结结束缝合完成肋间肌及壁层胸膜的缝合。
  Arms: Experimental group

SUMMARY:
The purpose of this trial is to understand whether intercostal suture can effectively prevent postoperative chest wall lung herniation, mainly to verify the following questions Can intercostal suture reduce postoperative chest wall lung herniation The hemostatic effect and hemostatic time of intercostal suture on intercostal muscle incision bleeding during surgery The researchers will divide the participants into two groups, one group will receive intercostal suture, and the other group will not receive intercostal suture, that is, conventional suture The participants will Receive or not receive intercostal suture during surgery Hemostatic effect and hemostasis time of rib intermuscular incision bleeding during surgery Chest CT will be reviewed 3 months after surgery to observe the chest wall incision

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lung resection via multiport thoracoscopic surgery
* Age greater than or equal to 18 years
* No history of thoracic surgery

Exclusion Criteria:

* Be converted to a thoracoscopic-assisted mini-thoracotomy,a rib retractor becomes necessary.
* Be converted to thoracotomy or a conventional posterolateral incision may be necessary based on the specific intraoperative circumstances.
* Uniportal thoracoscopic surgery
* History of ipsilateral thoracic surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 104 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Postoperative chest CT at 3 months | From enrollment to the end of treatment at 3 months
  Postoperative follow-up chest CT:If the CT indicates that the lung tissue at the main incision site has herniated through the intercostal space to the outside of the rib bony structure,it is considered positive;otherwise,it is negative.
Hemostasis time | From enrollment to the end of surgery
  Record the bleeding condition at the intercostal incision. If there is bleeding at the intercostal incision, record the hemostasis time in detail.

SECONDARY OUTCOMES:
Postoperative drainage volume within 3 days | Postoperative Day 1,Day 2,Day 3
  Record the volume of closed thoracic drainage every 24 hours,and document for 3 days postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR